CLINICAL TRIAL: NCT01410799
Title: Three Month Treatment of GHRH (Growth Hormone Releasing Hormone) in the Elderly
Brief Title: Three Month Treatment of Growth Hormone Releasing Hormone (GHRH) in the Elderly
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding ended
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 813246; P01AG000599 (NIH)
Record Dates: First submitted 2011-06-17; First posted 2011-08-05 (Estimated); Results first posted 2019-05-24 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Hormone Deficiency; Aging
Keywords: Growth Hormone Releasing Hormone; Growth Hormone Insufficiency; Aging; Growth Hormone; Physiologic Effects of Drugs; Hormones, Hormone Substitutes, and Hormone Antagonists; Hormones
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Growth Hormone-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Growth Hormone Releasing Hormone (GHRH) (Experimental): Drug: GHRH
  Interventions: Drug: Growth Hormone Releasing Hormone (GHRH )

INTERVENTIONS:
Drug: Growth Hormone Releasing Hormone (GHRH ) — GHRH administered subcutaneously at 2.0 mg/kg/dose bolus each night at 11:00 PM, 1:00 AM, 3:00 AM, and 5:00 AM for 12 weeks
  Other Names: Growth Hormone Releasing Factor

SUMMARY:
The purpose of the study is to evaluate the effect of a naturally occurring hormone, called Growth Hormone Releasing Hormone (GHRH) on the muscle, bone, and fat tissues of the body. GHRH stimulates the production of growth hormone (GH), which regulates the build up of many tissues in the body, including muscles and bones. Many elderly people have low levels of GH. The overall goal of this research is to determine the efficacy of GHRH to raise levels of GH and improve these body tissues. Healthy men and women age 65 and older will receive GHRH in four doses nightly for 12 weeks and assessed for changes in muscle strength, body mass, physical performance, and how the body uses sugar.

DETAILED DESCRIPTION:
Although multiple factors appear to be associated with the functional deterioration of advanced age, decreases in muscle mass and strength (sarcopenia) are commonly seen in aging subjects and are major risk factors for subsequent disability. There are many potential causes of sarcopenia and functional impairment in the elderly, including medical conditions such as cardiovascular disease, altered mood, and sedentary lifestyle. Hyposomatotropism, or decreased activity of growth hormone (GH), is one factor that has been implicated.

GH is a major anabolic hormone that exerts important stimulatory effects on protein synthesis. Many of the peripheral tissue effects of GH are mediated by insulin-like growth factor 1 (IGF-1) produced systemically by the liver or locally in tissues in response to GH stimulation. IGF-1, in turn, regulates GH secretion by negative feedback mechanisms at the pituitary gland. Several investigators have shown that aging is associated with a decrease in spontaneous GH secretion and IGF-1 levels. GH levels decline by 14% for each decade after puberty. Reduction of GH release in aging is thought to be associated with an increase in somatostatin tone, decrease in hypothalmic GHRH output, and diminished response to GHRH. The fact that aging is accompanied by a decrease in protein synthesis leading to a loss of lean body mass and a gain in body fat suggests that a decrease in GH secretion may contribute to these changes. It has been hypothesized that restoration of GH level in the elderly to the levels observed in younger individuals may lead to improvements in body composition. GH may also increase slow wave (delta or deep) sleep in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age of 65 years or older
* Fasting IGF-1 level <135ng/ml
* BMI 23-40 kg/m2
* Capable of giving informed consent

Exclusion Criteria:

* Diabetes mellitus or use of hypoglycemic agents
* Known coronary artery disease
* Liver disease, abnormal liver function tests (LRTs>2x upper limit of normal) or inflammatory bowel disease
* Renal insufficiency (serum creatinine > or = to 1.4 mg/dL)
* Hematocrit < 33% or > 50%
* History of malignancy < 5 years other than basal cell of the skin
* Chronic pulmonary disease or other systemic disorders which affect glucose hemostasis
* Use of growth hormone, corticosteroids, thiazide diuretics, estrogen supplements or androgen supplements
* Inability to perform strength or performance testing
* Uncontrolled hypertension (blood pressure >160/95
* NYHA Class III or IV heart failure
* Current smoking
* Alcohol use > or = to 30g/day
* Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study
* Participation in an investigational drug study within 6 weeks prior to screening visit
* Plan to change diet or exercise regimen during the study period

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dariush Elahi, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania-UPHS Presbyterian Campus, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Growth Hormone Releasing Hormone (GHRH)
Started | 13
Completed | 0
Not Completed | 13
Not completed — PI decision | 13

BASELINE CHARACTERISTICS:
Arm/Group | Growth Hormone Releasing Hormone (GHRH)
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 13
Sex/Gender, Customized [Count of Participants; unit: Participants] — N/A. Documents unavailable to determine number of males and number of females. Study was terminated before any outcome data were collected.
  Participants
    Male or Female | NA — N/A. Documents unavailable to determine number of males and number of females. Study was terminated before any outcome data were collected.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Muscle Strength
Description: Pre-drug and post-drug 1 RM (Repetition Maximum) testing
Time Frame: 12 weeks
Population: Study was terminated, no data collected.
Arm/Group | Growth Hormone Releasing Hormone (GHRH)
Number analyzed (Participants) | 0

2. Secondary Outcome: Glucose Homeostasis
Description: Glucose clamp study at week 12 of study drug use
Time Frame: 12 weeks
Population: Study was terminated, no data collected.
Arm/Group | Growth Hormone Releasing Hormone (GHRH)
Number analyzed (Participants) | 0

3. Secondary Outcome: Fat-free and Lean Mass
Description: iDXA scan
Time Frame: baseline and 12 weeks
Population: Study was terminated, no data collected.
Arm/Group | Growth Hormone Releasing Hormone (GHRH)
Number analyzed (Participants) | 0

4. Secondary Outcome: Fuel Utilization
Description: Assessment of resting metabolic rate
Time Frame: baseline and 12 weeks
Population: Study was terminated, no data collected.
Arm/Group | Growth Hormone Releasing Hormone (GHRH)
Number analyzed (Participants) | 0

5. Secondary Outcome: Physical Performance
Description: 6 Minute Walk Test
Time Frame: Baseline and 12 weeks
Population: Study was terminated, no data collected.
Arm/Group | Growth Hormone Releasing Hormone (GHRH)
Number analyzed (Participants) | 0

6. Secondary Outcome: Tolerability of Nocturnal Administration
Description: Subjects record diary of drug administration in evening and morning describing any issues with pump system for drug delivery, local skin issues at site of injection or other adverse events. Study nurses also record telephone contact with subjects every other day for first week of dosing and weekly for first month.
Time Frame: Ongoing throughout 12 weeks
Population: Study was terminated, no data collected.
Arm/Group | Growth Hormone Releasing Hormone (GHRH)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Growth Hormone Releasing Hormone (GHRH)
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 1/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Growth Hormone Releasing Hormone (GHRH) (N=13)
Fatigue (Endocrine disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes